CLINICAL TRIAL: NCT00460213
Title: Study on Optimal Anti-hypertensive Therapy With Valsartan by Using Home Blood Pressure Measurement
Brief Title: Valsartan Optimal Therapy Against Elevated Home Blood Pressure Research（VOYAGER）Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kitakyushu-Tsuyazaki Hospital (Other)
Responsible Party: Principal Investigator, Koshiro Fukiyama, Honorary Director, Kitakyushu-Tsuyazaki Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KIT-061003-1; ISRCTN1150
Record Dates: First submitted 2007-03-28; First posted 2007-04-13 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
Keywords: home blood pressure
MeSH Terms: conditions — Hypertension | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valsartan (Experimental)
  Interventions: Drug: Valsartan 80mg daily; Drug: Valsartan 160mg daily

INTERVENTIONS:
Drug: Valsartan 80mg daily
Drug: Valsartan 160mg daily

SUMMARY:
The purpose of this study is to compare improvement percentage of urinary albumin excretion between valsartan 80 mg- and valsartan 160 mg-based therapy in patient with morning hypertension.

DETAILED DESCRIPTION:
The cardiovascular diseases such as stroke and myocardial infarction consist 50% of the cause of death in Japanese population. Numerous mega trials have shown that strict anti-hypertensive therapy could reduce cardiovascular morbidity and mortality in hypertensive patients.

It is reported, however, over 50% hypertensive patients have not been controlled below therapeutic target blood pressure that the JSH2004 guideline recommends.

Recently use of Angiotensin II receptor blockers (ARBs) is increasing progressively for their pharmacological action on organ protection as well as potent reduction in blood pressure. However, usual dosage of ARB in Japan is almost half of that in the mega trials executed in Europe and America. Lower dosage compared to western countries might be a reason why cardiovascular events are not fully reduced in Japan.

Valsartan optimal therapy against elevated home blood pressure research (VOYAGER) study will be a multi-center, open-label, randomized, active-controlled study to evaluate the following; improvement percentage of urinary albumin exception, home blood pressure, hospital blood pressure, incidence of stroke, cardiovascular disease, and microangiopathy with valsartan 80 mg- or valsartan 160 mg based therapy in patients with elevated morning home blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged over 20 years and less than 80 years, regardless of sex.
* Patients with stable seated morning home blood pressure of over 135 mmHg and/or diastolic blood pressure of over 85 mmHg within 1 to 2 weeks.
* Patients who are on therapy with conventional dosage of ARB.

Exclusion Criteria:

* Patients who are difficult to measure home blood pressure.
* Patients with secondary hypertension or malignant hypertension.
* Patients with seated systolic blood pressure of over 200 mmHg.
* Patients with seated diastolic blood pressure of over 120 mmHg.
* Patients with a history of cerebrovascular disorder or myocardial infarction or heart failure within 6 months prior to enrolment in the study.
* Patients with atrial fibrillation, atrial flutter, or serious arrhythmia.
* Patients with renal dysfunction with serum creatinine level of over 2 mg/dL.
* Patients with serious liver dysfunction.
* Patient with HbA1C of over 8 percent.
* Patient with positive albuminuria by dip and read stick test.
* Patient treated with any angiotensin converting enzyme inhibitor
* Pregnant women
* Patients with a history of hypersensitivity to valsartan.
* Other patients who are judged to be inappropriate for the study by the investigator or sub-investigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Improvement percentage of urinary albumin excretion | 3, 6, 9, and 12 months

SECONDARY OUTCOMES:
home blood pressure; hospital blood pressure; stroke; cardiovascular disease; microangiopathy | every month

CONTACTS AND LOCATIONS:
Overall Officials: Koshiro Fukiyama, MD, Study Chair — Japan Seamen's Relief Association Moji Hospital
Locations (1):
- Koshiro Fukiyama, Kitakyushu, Fukuoka, Japan